CLINICAL TRIAL: NCT01087619
Title: Primary Hyperparathyroidism in Patients Older Than 65 Years: A Prospective Randomized Trial of Surgical Treatment Compared With Follow-up
Brief Title: Surgery for Primary Hyperparathyroidism (pHPT) in Patients Older Than 65 Years Compared With Follow-up
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/51
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Primary Hyperparathyroidism
Keywords: Hyperparathyroidism, primary; Aged 66 years or older; Mild hypercalcaemia; Surgical Procedures, Elective; Indication; Osteoporosis; Cognitive function; Atherosclerosis; Follow-up; Randomized trial
MeSH Terms: conditions — Hyperparathyroidism, Primary; Osteoporosis; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up (No Intervention): Patients diagnosed biochemically and clinically with primary hyperparathyroidism who are followed only
- Surgery (Experimental): Patients diagnosed biochemically and clinically with primary hyperparathyroidism who are treated with parathyroid surgery
  Interventions: Procedure: Parathyroid surgery

INTERVENTIONS:
Procedure: Parathyroid surgery — Parathyroid Surgery (regardless of surgical strategy; i.e., focused operation, unilateral- or bilateral neck exploration)
  Other Names: BA
  Arms: Surgery

SUMMARY:
General consensus and contemporary guidelines, recommend surgery for primary hyperparathyroidism (pHPT)for all patients below the age of 50, for patients with pronounced hypercalcemia and for patients with organ complications to the disease (osteoporosis and decreased renal function).

The purpose of this study is to determine if surgery for pHPT, is appropriate for patients with moderate to mild hypercalcemia older than 65 years of age.

The hypothesis of the study is that surgery for pHPT in patients older than 65 years of age, and with mild hypercalcemia, will increase bone density and hence decrease future risk for fragility fractures compared to patients with follow-up only.

DETAILED DESCRIPTION:
The majority of patients diagnosed and operated due to primary HPT in Scandinavia are older than 65 years of age. The vast majority of the patients have mild aberrations of serum calcium (< 1.50 mmol/l ionized calcium), and some patients may even be asymptomatic. The present trial is designed to clarify the indications for surgical treatment in this large subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary Hyperparathyroidism
* No previous parathyroid surgery
* Sporadic disease

Exclusion Criteria:

* Z-score of Bone density < -2.5 SD (regardless of site)
* Serum level of ionized calcium > 1.50 mmol/L
* Inability to understand given information or to comply with scheduled follow-up
* Symptoms of hypercalcaemia for which specific medical treatment has been prescribed

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone density at the hip | At two years
  Bone density is assessed with DEXA (dual energy x-ray absorptiometry), at the hip.

SECONDARY OUTCOMES:
Bone density at the lumbar spine | At two years
  Bone density is assessed with DEXA (dual energy x-ray absorptiometry) at the lumber spine
Blood lipids | At two years
  Triglyceride and cholesterol concentrations of whole serum and of the lipoprotein classes; low-density-lipoprotein (LDL), very-low-density-lipoprotein (VLDL) and high-density-lipoprotein (HDL).
Cardiac function | At two years
  Cardiac function assessed with echocardiography; Left ventricular ejection fraction (EF), Left ventricular end-diastolic diameter (LVDD), Left ventricular mass index (LVMI), Ratio between mitral peak velocity flow of the early filling wave and the atrial filling wave (E/A ratio).
Cognitive function | At two years
  Mini Mental State Examination test (MMSE), for cognitive function.
  A Quich Test (AQT), for cognitive speed
Atherosclerosis | At one two years
  Carotid ultrasound/duplex scans with evaluation of intimal-medial thickness and plaques.
Oral glucose tolerance | At two years
  Oral glucose tolerance test (75 Gram), with measurement of blood glucose and insulin after 60, 120 and 180 min.
Blood pressure (systolic and diastolic) | At two years
  24 hours blood pressure measurement
Renal function | At two years
  GFR measured by the clearance of iohexol and urinary albumin excretion

CONTACTS AND LOCATIONS:
Overall Officials: Anders OJ Bergenfelz, MD, PhD, Principal Investigator — Skåne University Hospital, Department of Surgery, Lund
Locations (1):
- Skåne University Hospital, Department of Surgery, Lund, Lund, Sweden